CLINICAL TRIAL: NCT01203475
Title: Growth Observational Study
Acronym: Growth
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Richard A. Ehrenkranz/ Lead Principal Investigator, Yale University
Other Study IDs: NICHD-NRN-0013; U10HD021364 (NIH); U10HD027853 (NIH); M01RR008084 (NIH); U10HD027851 (NIH); U01HD019897 (NIH); U10HD027856 (NIH); M01RR000750 (NIH); U10HD021397 (NIH); U10HD027881 (NIH); M01RR000997 (NIH); U10HD027880 (NIH); M01RR000070 (NIH); U10HD021415 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027904 (NIH); U10HD027871 (NIH); M01RR006022 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Growth Curve; Head Circumference; Length
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study was a multicenter, prospective cohort study to define postnatal longitudinal growth for very low birth weight (VLBW) infants. The objectives were: 1) to develop postnatal growth curves for VLBW preterm infants that would permit an assessment of growth velocity; 2) to relate growth velocity and nutritional practices (duration of parenteral nutrition, age at first enteral feeding, and age at full enteral feeding); 3) to compare growth velocity in infants who are small-for-gestational age (SGA) with infants who are appropriate-for-gestational age (AGA); and 4) to relate growth velocity to several common, major morbidities, including chronic lung disease (CLD), nosocomial infection (or late-onset infection) and necrotizing enterocolitis (NEC). These growth data may be useful in identifying preterm infants who are growing slowly despite current nutritional support and in designing and performing clinical trials of nutritional interventions.

DETAILED DESCRIPTION:
Previous growth curves for premature infants were based on a 1948 study of 100 infants. More recent reports described growth rates for VLBW infants exceeded those predicted by the previous study. The authors suggested that the differences may reflect changes in nutritional management and cautioned that the observed growth rates may not be optimal. Although a greater number of extremely low birth weight infants were included in these studies, data for infants with birth weights <750 g was still limited.

This study was a multicenter, prospective cohort study to define postnatal longitudinal growth for very low birth weight (VLBW) infants. The objectives were: 1) to develop postnatal growth curves for VLBW preterm infants that would permit an assessment of growth velocity; 2) to relate growth velocity and nutritional practices (duration of parenteral nutrition, age at first enteral feeding, and age at full enteral feeding); 3) to compare growth velocity in infants who are small-for-gestational age (SGA) with infants who are appropriate-for-gestational age (AGA); and 4) to relate growth velocity to several common, major morbidities, including chronic lung disease (CLD), nosocomial infection (or late-onset infection) and necrotizing enterocolitis (NEC). These growth data may be useful in identifying preterm infants who are growing slowly despite current nutritional support and in designing and performing clinical trials of nutritional interventions.

Data were collected on 1660 infants with birth weights between 501 to 1500 g who were inborn or admitted at 24 hours of age or less to 1 of the 12 National Institute of Child Health and Human Development (NICHD) Neonatal Research Network centers between August 31, 1994 and August 9, 1995, survived >7 days (168 hours) and were free of major congenital anomalies. Infants were weighed daily for a minimum of 14 days or until birth weight was regained, whichever occurred later, and then weekly. Recumbent length was measured weekly with a Premie Length Board. Head circumference (HC) was measured weekly. Midarm circumference (MAC) was measured weekly. Length, HC, and MAC measurements were each performed twice.

ELIGIBILITY:
Inclusion Criteria:

* Infants with birth weights between 501 to 1500g who were inborn or admitted at 24 hours of age or less
* Survived >7 days (168 hours)

Exclusion Criteria:

* Major congenital anomalies

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature infants born at NICHD Neonatal Research Network centers during the study period.
Sampling Method: Probability Sample
Enrollment: 1660 (Actual)
Dates: Start 1994-08; Primary Completion 1995-08 (Actual); Study Completion 1995-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Ehrenkranz, MD, Study Director — Yale University; Avroy A. Fanaroff, MD, Principal Investigator — Case Wester Reserve University; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Barbara J. Stoll, MD, Principal Investigator — Emory University; Joel Verter, PhD, Principal Investigator — George Washington University; James A. Lemons, MD, Principal Investigator — Indiana University; Charles R. Bauer, MD, Principal Investigator — University of Miami; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; David K. Stevenson, MD, Principal Investigator — Stanford University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee at Memphis; Jon E. Tyson, MD, Principal Investigator — University of Texas; Seetha Shankaran, MD, Principal Investigator — Wayne State University; William Oh, MD, Principal Investigator — Brown University, Womens and Infants Hospital
Locations (13):
- United States (13):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Background] Dusick AM, Poindexter BB, Ehrenkranz RA, Lemons JA. Growth failure in the preterm infant: can we catch up? Semin Perinatol. 2003 Aug;27(4):302-10. doi: 10.1016/s0146-0005(03)00044-2. PMID 14510321
- [Result] Ehrenkranz RA, Younes N, Lemons JA, Fanaroff AA, Donovan EF, Wright LL, Katsikiotis V, Tyson JE, Oh W, Shankaran S, Bauer CR, Korones SB, Stoll BJ, Stevenson DK, Papile LA. Longitudinal growth of hospitalized very low birth weight infants. Pediatrics. 1999 Aug;104(2 Pt 1):280-9. doi: 10.1542/peds.104.2.280. PMID 10429008
- [Result] Ehrenkranz RA, Dusick AM, Vohr BR, Wright LL, Wrage LA, Poole WK. Growth in the neonatal intensive care unit influences neurodevelopmental and growth outcomes of extremely low birth weight infants. Pediatrics. 2006 Apr;117(4):1253-61. doi: 10.1542/peds.2005-1368. PMID 16585322
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/